CLINICAL TRIAL: NCT05302167
Title: Feasibility Study of an Adapted App-based Anxiety Intervention ('Molehill Mountain') for Autistic People.
Brief Title: Molehill Mountain Feasibility Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1286908
Record Dates: First submitted 2022-02-04; First posted 2022-03-31 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Autism
MeSH Terms: conditions — Anxiety Disorders; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility/ acceptability (Experimental)
  Interventions: Behavioral: Molehill Mountain app; Device: Molehill Mountain app

INTERVENTIONS:
Behavioral: Molehill Mountain app — The Molehill Mountain app (currently Version 2) was developed jointly by King's College London (Lead: Prof Emily Simonoff; Advisors: Dr Ann Ozsivadjian and Dr Rachel Kent) and UK autism charity Autistica (Product Owner: Andy Clarke; Product Designer: Joanna Alpe) for use by autistic people aged ≥12-years (https://www.autistica.org.uk/molehill-mountain).
  The app was designed based on a self-guided paper-and-pencil CBT toolkit adapted for autism by Professor Emily Simonoff. Since the first version of Molehill Mountain (a two-week long programme) was launched in 2016, and based on surveys of autistic people and five rounds of prototype testing, the Molehill Mountain V2 app was relaunched in April 2021 as a three-month long app-based programme with enhanced interactive features. This 3-month V2 Molehill Mountain app, with enhanced interactive features supporting short daily logins, that will be implemented in the current study.
Device: Molehill Mountain app — As above.

SUMMARY:
Up to half of autistic people experience anxiety symptoms, which can have a significant impact on everyday wellbeing. However, there are currently very few effective, evidence-based interventions to support autistic people in managing anxiety; and many autistic people face barriers in accessing inperson health and social care services. Therefore, developing new interventions (and/ or adapting existing ones) that improve anxiety, in a way that meets the needs of autistic people, represents the autism community's number one priority for research and clinical practice.

Addressing this priority, the investigators will test the acceptability and feasibility of a new, app-based therapeutic approach for anxiety ('Molehill Mountain') that has been developed with, and adapted for, autistic people aged 12-years and over using adapted Cognitive Behavioural therapy principles. This means that information will be collected from autistic people accessing clinical services on whether they would choose to use the anxiety app, whether the app is simple to administer and use, how it is used, how it can be improved, and whether it is effective in reducing anxiety symptoms and/ or enhancing other outcomes, such as everyday wellbeing and functioning.

The evidence from this project will inform the future optimisation and implementation of Molehill Mountain in a randomised-controlled trial, with the ultimate aim of transforming long-term healthcare delivery for autistic people.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16-years.
* Autism diagnosis.
* Current mild-to-severe anxiety symptom severity, as assessed at screening (and currently in touch with mental health services e.g., referred, on the waitlist).
* Able and willing to provide verbal and written informed consent to take part in the study.
* Access to Molehill Mountain app via SmartPhone or other Smart device.

Exclusion Criteria:

* Difficulties with reading/ writing to the extent that the app is inaccessible.
* High risk of self-harm that make participation in the study inappropriate for the individual's current level of clinical need (as assessed by clinical team).
* Attended ≥ 6 sessions of individual or group therapy (e.g., cognitive behavioural therapy) in the past 6-months, which would make it impossible to parse out the effects of the app from existing therapy.
* If using psychotropic medication, this medication/ dose must have been stable for a minimum of 8-weeks on entry to the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Change in 7-item Generalised Anxiety Disorder Scale (GAD-7) | Week 0 (+/-2); Week 13 (+/-2); Week 24 (+/- 4); Week 32 (+/-4); Week 41 (+/-4)
  Minimum score = 0; Maximum score = 21; Higher scores indicate more severe anxiety.
App acceptability/ feasibility survey | Week 13 (+/-2)
  A survey developed by the investigator team to assess the acceptability and feasibility of Molehill Mountain app use by autistic adolescents/ adults in a clinically derived sample. Key indices incorporated in post-study app use experience surveys include: 1) the preparedness of participants to be randomised in a future trial; 2) ease of app administration and use; 3) preferred app features, content, and structure; 4) non-preferred app features, content, and structure; 5) experiences of app technical functionality; and 6) subjective reflections on the impact of app use on anxiety and everyday wellbeing/ functioning.

SECONDARY OUTCOMES:
Change in Medication/ service use | Week 0 (+/-2); Week 13 (+/-2); Week 24 (+/- 4); Week 32 (+/-4); Week 41 (+/-4)
  To indicate changes in medication (number of medications, dose, frequency) and/ or clinical service use (number of appointments, attendance, length of engagement with services) with using the Molehill Mountain app to manage anxiety.
Change in Goal Attainment Scaling | Week 0 (+/-2); Week 13 (+/-2); Week 24 (+/- 4); Week 32 (+/-4); Week 41 (+/-4)
  Participants will choose 3 priority goals from a list of functional outcomes, including feeling less anxious, understanding anxiety better, understanding anxiety triggers better, and reducing anxiety across key areas of everyday life (e.g., relationships, social encounters, communication, school/ work, leisure, sensory). Participants will rate their progress in relation to these 3 goals on a scale from 1 (a very long way from this goal) to 7 (achieved this goal).

CONTACTS AND LOCATIONS:
Overall Officials: Emily Simonoff, MD; PhD, Principal Investigator — King's College London; Declan Murphy, MD; PhD, Principal Investigator — MD; PhD
Locations (2):
- United Kingdom (2):
  - King's College London, London
  - South London and Maudsley NHS Foundation Trust (SLaM), London

IPD SHARING:
Plan to Share IPD: Yes
The research team will produce a fully anonymised (i.e., no longer coded, or including any identifiable or special category data) quantitative dataset at the end of the study that will be openly accessible. Participant consent will be gained to do so.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The dataset will become available at the end of the study (estimated March 2023). Due to its fully anonymised nature, this dataset will be available indefinitely.

REFERENCES:
- [Derived] Oakley B, Boatman CA, Baldoza S, Hearn A, Larkworthy C, Kent R, Ozsivadjian A, Doswell S, Dittner A, Roestorf A, Rawal D, Carter B, Simonoff E; Molehill Mountain Advisory Group. Feasibility Study of a Novel App-Based Anxiety Intervention for Autistic People. Autism Res. 2025 Dec 14. doi: 10.1002/aur.70153. Online ahead of print. PMID 41392571
- [Derived] Oakley B, Boatman C, Doswell S, Dittner A, Clarke A, Ozsivadjian A, Kent R, Judd A, Baldoza S, Hearn A, Murphy D, Simonoff E; Molehill Mountain Advisory Group. Molehill Mountain feasibility study: Protocol for a non-randomised pilot trial of a novel app-based anxiety intervention for autistic people. PLoS One. 2023 Jul 5;18(7):e0286792. doi: 10.1371/journal.pone.0286792. eCollection 2023. PMID 37406026

DOCUMENTS (1):
  • Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT05302167/ICF_000.pdf